CLINICAL TRIAL: NCT06885541
Title: Detection of Internal Tremors by Oscillometry in Parkinson's Patient : a Pilot Study
Brief Title: Detection of Internal Tremors by Oscillometry in Parkinson's Patient
Acronym: TREMOS-PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/25/0028; 2025-A00133-46 (Other: ANSM)
Record Dates: First submitted 2025-02-27; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Internal tremor; Tremor; Wearable devices; Accelerometer; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Tremor

STUDY DESIGN:
Intervention Model Description: Two groups of participants : the first group consists of Parkinson's disease patients in the off phase, while the second group consists of healthy participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's disease patients (Other): Parkinson's disease patient in the off phase.
  Interventions: Diagnostic Test: Detection of objective internal tremors
- Healthy participants (Other): Healthy participants
  Interventions: Diagnostic Test: Detection of objective internal tremors

INTERVENTIONS:
Diagnostic Test: Detection of objective internal tremors — head-mounted motion sensors

SUMMARY:
The goal of the present study is to objectively access the presence of an Internal Tremor in Parkinson's disease. Inertial sensors will be used to detect the presence of a rhythmic oscillation of 3-4 Hz. The study will be performed in both Parkinson's disease patients and healthy controls to ascertain the specificity of this type of tremor.

DETAILED DESCRIPTION:
The interest in finding prodromal symptoms in Parkinson's disease has been growing. Internal tremor, felt subjectively by the patients, have been reported in some studies as being present on the Prodromal phases of the disease. An objective identification of this tremor has never been made. In this study we propose to objectively access the presence of Internal Tremor in Parkinson's Disease patients using accelerometers. A control population of healthy subjects will also be evaluated to confirm the specificity of tremor for a PD population.

ELIGIBILITY:
Inclusion Criteria:

(For the experimental group)

* Patient with idiopathic parkinson's disease
* Mini Mental State Evaluation score above or equal to 25
* Hoehn and Yahr scale score of ≤3 in the OFF phase, with postural stability allowing the patient to stand unaided for 1 minute.
* Able to walk unassisted
* No major osteoarticular issues
* Presence of another neurological condition that may affect gait
* Willing to undergo accelerometry in the OFF state

(For the control group)

* Healthy volunteer subjects matched for age (+/- 5 years) and sex
* Mini Mental State Evaluation score above or equal to 25

Exclusion Criteria:

(For the experimental group)

* Patients with an atypical parkinsonian syndrome
* Patients unable to walk or stand for more than one minute in the off state
* Parkinson's patients treated with deep brain stimulation, apomorphine pump, or duodopa intestinal infusion, and foslevodopa
* Pregnant patients

(For the control group)

* Participants with significant gait impairment (osteoarticular disorder)
* Those with a neurological disease that, in the investigator's judgment, may interfere with the study's outcome measure
* Participants with a clinical tremor that may interfere with the measurement of the primary outcome (e.g., essential tremor, thyroid disease, or tremors induced by medication)
* Pregnant participants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Difference in intensity of the peak power at 4-6 Hz | Baseline
  Difference in maximum signal power in the 4 to 6 Hz frequency band of the objective internal tremor, recorded from the head sensor, between the group of Parkinson's patients and a matched group of healthy volunteers.

SECONDARY OUTCOMES:
Association between subjective internal tremors and frequency peak between 4 and 6 Hz | Baseline
  The difference between objective internal tremor and subjective internal tremor is a descriptive outcome measure and will be assessed using the correlation coefficient between the score on the Internal Tremor Questionnaire, which measures subjective internal tremor intensity, and the maximum signal power in the 4 to 6 Hz frequency band of objective internal tremor.
  The Internal Tremor Questionnaire measures the intensity of internal tremor perceived by subjects. It consists of 13 questions. At the end of the questionnaire, the patient receives a score out of 13, with 0 being the best score and 13 being the worst score.
  The objective internal tremor is measured via the sensors measure the movement associated with muscle contractions. The data is recorded as a time series, which represents the tremor amplitude at discrete time intervals.
Association between Objective Internal Tremor and Motor Symptom Severity in Parkinson's Disease as Assessed by the MDS-UPDRS | Baseline
  The association between objective internal tremor and symptom severity will be a descriptive analyses and assessed using the correlation coefficient between the score on the MDS-UPDRS (Part III - Motor Symptoms), which evaluates motor symptom severity in Parkinson's patients, and the maximum signal power in the 4 to 6 Hz frequency band of objective internal tremor.
  The scale is a composite, with scores ranging from 0 to 120, where higher scores indicate greater symptom severity, meaning that a lower score reflects a better clinical condition.
  see above for how the Objective Internal tremor is assessed.
Evaluation of Objective Internal Tremor Powers Detected by Different Sensors in Parkinson's Disease | Baseline
  The powers of the objective internal tremor detected by the other sensors will be assessed by comparing the maximum signal power in the 4 to 6 Hz frequency band of each sensor (back and thigh on the most affected side of Parkinson's disease) to the head sensor.
Evaluation of Acceptability of Motion Sensor Examination Using the Visual Analog Scale | Baseline
  Acceptability will be assessed using the scores from the Visual Analog Scale (VAS), (0 = not acceptable to 10 = completely acceptable), measuring the acceptability of the motion sensor examination in patients and controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Purpan Hospital, Toulouse, Occitanie, France

REFERENCES:
- [Background] Mendonca MD, Ferreira PC, Oliveira F, Barbosa R, Meira B, Costa DC, Oliveira-Maia AJ, da Silva JA. Relative sparing of dopaminergic terminals in the caudate nucleus is a feature of rest tremor in Parkinson's disease. NPJ Parkinsons Dis. 2024 Nov 18;10(1):209. doi: 10.1038/s41531-024-00818-8. PMID 39557871
- [Background] Schrag A, Bohlken J, Dammertz L, Teipel S, Hermann W, Akmatov MK, Batzing J, Holstiege J. Widening the Spectrum of Risk Factors, Comorbidities, and Prodromal Features of Parkinson Disease. JAMA Neurol. 2023 Feb 1;80(2):161-171. doi: 10.1001/jamaneurol.2022.3902. PMID 36342675
- [Background] Cochrane GD, Rizvi S, Abrantes A, Crabtree B, Cahill J, Friedman JH. Internal tremor in Parkinson's disease, multiple sclerosis, and essential tremor. Parkinsonism Relat Disord. 2015 Oct;21(10):1145-7. doi: 10.1016/j.parkreldis.2015.07.014. Epub 2015 Jul 18. PMID 26307481
- [Background] Shulman LM, Singer C, Bean JA, Weiner WJ. Internal tremor in patients with Parkinson's disease. Mov Disord. 1996 Jan;11(1):3-7. doi: 10.1002/mds.870110103. PMID 8771060
- [Background] Bhatia KP, Bain P, Bajaj N, Elble RJ, Hallett M, Louis ED, Raethjen J, Stamelou M, Testa CM, Deuschl G; Tremor Task Force of the International Parkinson and Movement Disorder Society. Consensus Statement on the classification of tremors. from the task force on tremor of the International Parkinson and Movement Disorder Society. Mov Disord. 2018 Jan;33(1):75-87. doi: 10.1002/mds.27121. Epub 2017 Nov 30. PMID 29193359
- [Background] Abusrair AH, Elsekaily W, Bohlega S. Tremor in Parkinson's Disease: From Pathophysiology to Advanced Therapies. Tremor Other Hyperkinet Mov (N Y). 2022 Sep 13;12:29. doi: 10.5334/tohm.712. eCollection 2022. PMID 36211804
- [Background] Poewe W, Seppi K, Tanner CM, Halliday GM, Brundin P, Volkmann J, Schrag AE, Lang AE. Parkinson disease. Nat Rev Dis Primers. 2017 Mar 23;3:17013. doi: 10.1038/nrdp.2017.13. PMID 28332488
- [Background] Jennings D, Siderowf A, Stern M, Seibyl J, Eberly S, Oakes D, Marek K; PARS Investigators. Conversion to Parkinson Disease in the PARS Hyposmic and Dopamine Transporter-Deficit Prodromal Cohort. JAMA Neurol. 2017 Aug 1;74(8):933-940. doi: 10.1001/jamaneurol.2017.0985. PMID 28595287
- [Background] Postuma RB, Iranzo A, Hu M, Hogl B, Boeve BF, Manni R, Oertel WH, Arnulf I, Ferini-Strambi L, Puligheddu M, Antelmi E, Cochen De Cock V, Arnaldi D, Mollenhauer B, Videnovic A, Sonka K, Jung KY, Kunz D, Dauvilliers Y, Provini F, Lewis SJ, Buskova J, Pavlova M, Heidbreder A, Montplaisir JY, Santamaria J, Barber TR, Stefani A, St Louis EK, Terzaghi M, Janzen A, Leu-Semenescu S, Plazzi G, Nobili F, Sixel-Doering F, Dusek P, Bes F, Cortelli P, Ehgoetz Martens K, Gagnon JF, Gaig C, Zucconi M, Trenkwalder C, Gan-Or Z, Lo C, Rolinski M, Mahlknecht P, Holzknecht E, Boeve AR, Teigen LN, Toscano G, Mayer G, Morbelli S, Dawson B, Pelletier A. Risk and predictors of dementia and parkinsonism in idiopathic REM sleep behaviour disorder: a multicentre study. Brain. 2019 Mar 1;142(3):744-759. doi: 10.1093/brain/awz030. PMID 30789229
- [Background] Mahlknecht P, Seppi K, Poewe W. The Concept of Prodromal Parkinson's Disease. J Parkinsons Dis. 2015;5(4):681-97. doi: 10.3233/JPD-150685. PMID 26485429
- [Background] Berg D, Postuma RB, Adler CH, Bloem BR, Chan P, Dubois B, Gasser T, Goetz CG, Halliday G, Joseph L, Lang AE, Liepelt-Scarfone I, Litvan I, Marek K, Obeso J, Oertel W, Olanow CW, Poewe W, Stern M, Deuschl G. MDS research criteria for prodromal Parkinson's disease. Mov Disord. 2015 Oct;30(12):1600-11. doi: 10.1002/mds.26431. PMID 26474317
- [Background] Berg D, Borghammer P, Fereshtehnejad SM, Heinzel S, Horsager J, Schaeffer E, Postuma RB. Prodromal Parkinson disease subtypes - key to understanding heterogeneity. Nat Rev Neurol. 2021 Jun;17(6):349-361. doi: 10.1038/s41582-021-00486-9. Epub 2021 Apr 20. PMID 33879872
- [Background] Heim B, Krismer F, De Marzi R, Seppi K. Magnetic resonance imaging for the diagnosis of Parkinson's disease. J Neural Transm (Vienna). 2017 Aug;124(8):915-964. doi: 10.1007/s00702-017-1717-8. Epub 2017 Apr 4. PMID 28378231
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] Dorsey ER, Sherer T, Okun MS, Bloem BR. The Emerging Evidence of the Parkinson Pandemic. J Parkinsons Dis. 2018;8(s1):S3-S8. doi: 10.3233/JPD-181474. PMID 30584159
- [Background] Bloem BR, Okun MS, Klein C. Parkinson's disease. Lancet. 2021 Jun 12;397(10291):2284-2303. doi: 10.1016/S0140-6736(21)00218-X. Epub 2021 Apr 10. PMID 33848468